CLINICAL TRIAL: NCT01365832
Title: CRP Evolution Pattern in CPAP Treated Obstructive Sleep Apnea Patients. Does Gender Play a Role?
Brief Title: Change in C-reactive Protein (CRP) in Men and Women With Sleep Apnea After Continuous Positive Airway Pressure (CPAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Sophia Schiza, University of Crete
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSACRP-02
Record Dates: First submitted 2011-05-17; First posted 2011-06-03 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure; Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep apnea (Experimental): Participants with Obstructive Sleep Apnea (OSA).This arm will undergo a pre-treatment blood draw, six months of Continuous Positive Airway Pressure (CPAP) to treat OSA, and a post-treatment blood draw 3 and 6 months later.
  Intervention: Procedure: Continuous Positive Airway Pressure (CPAP)
  Interventions: Procedure: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Procedure: Continuous Positive Airway Pressure (CPAP) — Continuous positive airway pressure (CPAP) is the gold standard for Obstructive Sleep Apnea (OSA) management. Subjects with OSA will be trained in the use of CPAP and will be instructed to use CPAP every night for 6 months. These subjects will then return for a post-treatment blood draw 3 and 6 months after the start of effective CPAP treatment
  Other Names: positive pressure ventilation

SUMMARY:
C-reactive protein (CRP) is directly implicated in atherogenesis and associated cardiovascular morbidity in patients with obstructive sleep apnea (OSA). Effective Continuous Positive Airway Pressure (CPAP) treatment has been shown to gradually decrease CRP levels and thus consequently improve disease-related cardiovascular morbidity. However, the influence of gender on the CRP evolution pattern has never been assessed before. The aim of our study was to investigate possible gender differences in CRP evolution in OSA patients 3 and 6 months after the start of effective CPAP treatment.

DETAILED DESCRIPTION:
OSA is an independent risk factor for a number of cardiovascular diseases. One important possible mechanism underlying cardiovascular disease in patients with OSA is systemic inflammation. CRP, an acute phase reactant secreted by the liver, is one of the most actively studied biomarkers of low-grade inflammation, and numerous studies have shown that higher CRP levels are associated with high mortality and morbidity due to cardiovascular disease in men and women. In patients with OSA, the question as to whether or not CRP levels are elevated is still under debate. Although continuous positive airway pressure (CPAP) is effective in the management of OSA, conflicting data also exist regarding the effects of CPAP on CRP levels. However, none of the existing studies assessed the influence of gender on the CRP evolution pattern. Therefore, the aim of this study was to investigate possible gender differences in CRP evolution in patients with moderate to severe OSA, free of medical comorbidities, 3 and 6 months after the start of effective CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with apnoea-hypopnoea index >15/h

Exclusion Criteria:

* chronic obstructive pulmonary disease
* diabetes mellitus
* coronary artery disease
* congestive heart failure
* chronic renal failure
* known dyslipidemia
* smoking history
* hypothyroidism
* chronic or recent infectious or inflammatory disease
* use of anti-inflammatory or antibiotic drugs, or statins.
* postmenopausal females on estrogen replacement therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in CRP in OSA patients, according to gender, 3 and 6 months after the start of effective CPAP treatment. | Day 1, Month 3 and Month 6 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sophia E Schiza, MD, PhD, Study Chair — University of Crete; Charalampos Mermigkis, MD, Study Director — Sleep Disorders Center, Pulmonary Department, 401 General Army Hospital, Athens, Greece; Izolde Bouloukaki, MD, PhD, Principal Investigator — University of Crete
Locations (1):
- Sleep Disorders Unit, Department of Thoracic Medicine, Medical School, University of Crete, Heraklion, Crete, Greece